CLINICAL TRIAL: NCT04068727
Title: Leveraging Evidence-based Practices for Ambulatory VTE and Other Patients to be Safe With Direct Oral Anticoagulants: LEAVE Safe With DOACs
Brief Title: LEAVE Safe With DOACs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alok Kapoor, Associate Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H00017891; 1R18HS02592401 (Other Grant/Funding Number: Agency for Healthcare Research and Quality (AHRQ))
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases; Venous Thromboembolism; Atrial Fibrillation; Bleeding; Stroke
MeSH Terms: conditions — Cardiovascular Diseases; Venous Thromboembolism; Atrial Fibrillation; Hemorrhage; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Clinical Pharmacist Intervention (Experimental)
  Interventions: Other: Clinical Pharmacist Intervention

INTERVENTIONS:
Other: Clinical Pharmacist Intervention — After randomization, the pharmacist calls patients to assess drug choice and dose. Staff distribute manufacturer coupons and help patients apply for medication payment assistance. Pharmacist discusses DOAC alternatives with prescribe and provides DOAC education by discussing potential adverse effects, medication interactions, alarm symptoms, and lab work. Staff mail educational materials. Pharmacist documents concerns in the electronic health record and messages prescriber about missing lab work. Patients share medication-related concerns. Patients are provided with a phone number for non-education calls to discuss their medications from 6 AM - 10 PM on any day. The pharmacist offers dose de-escalation instructions based on the DOAC prescription. The pharmacist advises the continuity provider on DOAC duration and monitoring. For follow-up/perioperative support, the pharmacist reviews and recommends lab monitoring and gives DOAC interruption/resumption recommendations.
  Other Names: Clinical Pharmacist Intervention Based on Checklist Endorsed by the AC Forum
  Arms: Clinical Pharmacist Intervention

SUMMARY:
Given the risks associated with direct oral anticoagulants (DOACs) and the lack of defined pathways for patients prescribed this class of medications, the study intervention has the potential for an enormous impact in preventing medication errors and improving the quality of care transition, patient knowledge, and adherence with DOAC therapy.

DETAILED DESCRIPTION:
Patients first treated with direct oral anticoagulants (DOACs) in an ambulatory setting are at an elevated risk for adverse drug events (ADEs) or potential ADEs from medication errors. An intervention that integrates clinical pharmacists, a pharmacy technician, and follows a checklist published by experts at the Anticoagulation Forum can prevent adverse outcomes. The Investigators propose research on the effectiveness, implementation, and dissemination for a care transition intervention that follows the checklist which includes evaluation for appropriateness of DOAC use, assistance with drug procurement, telephone access to an anticoagulation expert, and other best practice recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* New prescription of DOAC within 4 days of consent OR continued DOAC use for a patient with new episode of worsening thromboembolic or bleeding event within 4 days of consent or discharged from the hospital with DOAC prescription within 4 days of consent
* Fluency in English, Portuguese, or Spanish

Exclusion Criteria:

* Currently hospitalized with inpatient status (as opposed to observation status)
* Age < 18
* Prisoners
* Pregnant patients (medications are contraindicated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Number of Direct Oral Anticoagulant (DOAC)-Related Clinically Important Medication Errors | 90 Days Post Enrollment
  The number of preventable, ameliorable and potential Adverse Drug Events (ADEs) that physician reviewers attribute to Direct Oral Anticoagulant (DOAC) medication. Each DOAC related clinically important medication error is counted as a separate event, enabling patients to have multiple events consistent with the literature.

SECONDARY OUTCOMES:
Patient Knowledge regarding Anticoagulation and Venus Thromboembolism (VTE) using the Anticoagulation and Venus Thromboembolism (VTE) knowledge questionnaire | 90 Days Post Enrollment
  Patient knowledge regarding Anticoagulation and Venus Thromboembolism (VTE) will be evaluated using a modified version of a 22-item instrument previously developed and tested by the institution. This instrument assesses patients' knowledge of warning signs of bleeding and new VTE, interactions with other medications, and complications of VTE. A low score indicate a low level of knowledge and a high score indicates a high level of knowledge regarding anticoagulation and VTE.
Number of missed or extra doses to assess medication adherence | 90 Days Post Enrollment
  Patients are asked to to count out the number of remaining pills from the last filled prescription and provide the fill date, number of pills dispensed, the schedule prescribed (either once or twice a day depending on DOAC), and skipped doses for deliberate interruption to determine medication adherence with the number of missed or extra doses.
Medication Possession Ratio (MPR) to assess medication adherence | 90 Days Post Enrollment
  Medication adherence is measured with Medication Possession Ratio (MPR) which is the ratio between the time a patient had medication on hand, the time that a patient is eligible to have a medication on hand, and the time that a patient is covered by the medication. The MPR ratio will be calculated by using available pharmacy data.
Proportion of days covered (PDC) to assess medication adherence | 90 Days Post Enrollment
  Proportion of Days Covered (PDC) is the ratio between the time that a patient has a medication on hand, the time that a patient is eligible to have a medication on hand, and the time that a patient is covered by the medication. Medication adherence will be evaluated using the mean PDC using available pharmacy data.

CONTACTS AND LOCATIONS:
Overall Officials: Alok Kapoor, MD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapoor A, Patel P, Mbusa D, Pham T, Cicirale C, Tran W, Beavers C, Javed S, Wagner J, Swain D, Crawford S, Darling C, ItoFuKunaga M, McManus D, Mazor K, Gurwitz J. Multicomponent Pharmacist Intervention Did Not Reduce Clinically Important Medication Errors for Ambulatory Patients Initiating Direct Oral Anticoagulants. J Gen Intern Med. 2023 Dec;38(16):3526-3534. doi: 10.1007/s11606-023-08315-z. Epub 2023 Sep 27. PMID 37758967
- [Derived] Pham T, Patel P, Mbusa D, Kapoor A, Crawford S, Sadiq H, Rampam S, Wagner J, Gurwitz JH, Mazor KM. Impact of a pharmacist intervention on DOAC knowledge and satisfaction in ambulatory patients. J Thromb Thrombolysis. 2023 Feb;55(2):346-354. doi: 10.1007/s11239-022-02743-0. Epub 2022 Dec 12. PMID 36510110